CLINICAL TRIAL: NCT06364436
Title: The Effect of Distant Reiki Therapy on the Postpartum Fatigue and Depression Risk: A Randomized Controlled Trial
Brief Title: Distant Reiki Therapy on Postpartum Period Fatigue and Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aksaray University (Other)
Responsible Party: Principal Investigator, İlknur Gökşin, Assistant Professor, Aksaray University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AksarayU1
Record Dates: First submitted 2024-04-04; First posted 2024-04-15 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: PostPartum Depression
Keywords: Postpartum period; Nursing; Distant Reiki; Postpartum depression; Fatigue
MeSH Terms: conditions — Depression, Postpartum; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reiki Energy therapy (Experimental): The women in the intervention group were explained how to perform the Reiki application, and the appropriate time for Reiki was planned. Pretest data were obtained by sending the data collection form, VAS-F and EPDS Google form link to women's phones via WhatsApp application.Then, according to Usui Reiki, researchers with Reiki Stage II and Reiki Master & Teacher degrees applied Reiki to women for 30 minutes consecutively on the 13th, 14th, 20th and 21st postpartum days (in the second and third postpartum weeks). Before each Reiki application, a reminder message was sent to the women informing them that the application would begin, and they were asked to fill out the VAS-F and EPDS again on the 28th day (fourth week) and 56th day (eighth week) postpartum. During this process, women who did not fill out the scale forms were contacted via phone and SMS and were asked to fill out the forms, and those who did not fill out the forms were excluded from the study.
  Interventions: Behavioral: Reiki energy therapy
- Control (No Intervention): No intervention was made to the women in the control group during the research. Women in the control group were asked to fill out the introductory information form and VAS-F and EPDS on the 13th postpartum day, and the VAS-F and EPDS form links were sent to their phones via WhatsApp on the 28th and 56th days.

INTERVENTIONS:
Behavioral: Reiki energy therapy — In order to perform distance Reiki application, the practitioner must have completed Reiki II level training according to the Traditional Usui Reiki system and must be attuned by a person with a Usui Reiki Master and Teacher degree. With harmony, the energy channels in the individual's body are opened and the harmonious individual becomes a tool of universal healing energy.
  Arms: Reiki Energy therapy

SUMMARY:
This research was conducted to evaluate the effect of Reiki therapy applied to women in the postpartum period on the risk of fatigue and postpartum depression.

DETAILED DESCRIPTION:
The postpartum period is a process in which the reproductive organs return to their prenatal state during the six weeks after birth, physiological and anatomical changes as well as physical, social and emotional changes occur in the woman, and new roles and responsibilities are learned. Most of the problems seen in this period appear in the first days and continue for periods ranging from six weeks to a year. Risk factors such as hormonal changes seen in the postpartum period in women, having a first baby, stressful life events, insufficient social support and problems in relationships with the spouse cause sleep disruption and fatigue, and therefore can negatively affect the psychological health of the woman.

While many women easily adapt to the physiological, psychological and social changes that occur with pregnancy and birth, psychological problems at various levels occur in women who cannot adapt. One of the psychological problems that develop during this period is postpartum depression. Postpartum depression develops due to biological, psychological and socio-cultural factors, can be seen within the first year after birth, disrupts the health of the mother and the family, and is characterized by symptoms such as sadness, hopelessness, weight changes, chronic fatigue, feelings of worthlessness or guilt, and difficulty in thinking and concentrating. It is a mental illness that is serious and requires treatment. When symptoms of fatigue and depression in the postpartum period are not noticed early and the woman is not provided with the support she needs, this makes it difficult for women to adapt to the postpartum period.

According to the holistic care philosophy, which has an important place in nursing and accepts that the whole is more than the sum of its parts, nurses should handle the individuals they care for with a holistic approach that includes physical health as well as emotional, mental and spiritual well-being. For this reason, in addition to pharmacological methods applied to reduce the fatigue levels of women in the postpartum period and reduce the risk of depression, complementary and alternative therapy methods such as massage, listening to music, acupressure, relaxation exercises and Reiki are also used in nursing research. Reiki, one of these alternative therapy methods, is based on the principle that a blockage or congestion in one of the energy centers such as the head, neck, chest, abdominal cavity and groin causes physical and psychological disorders. Reiki, a Japanese word, means life energy that exists everywhere. Reiki therapy has been defined as a complementary health approach in which the practitioner places his/her hands on or just above a person to direct universal energy to the receiving individual. Reiki, one of the healing methods based on life energy, is increasingly used in nursing studies. In studies conducted in the field of women's health in the literature; It has been determined that Reiki applied to female patients undergoing outpatient surgery before the operation reduces heart rate, systolic blood pressure and anxiety levels and reduces pain and analgesic use after abdominal hysterectomy. In studies conducted on the use of Reiki therapy in the postpartum period, Reiki applied to the post-cesarean intervention group on the first and second post-operative days reduced pain intensity, analgesic need and anxiety level, but had no effect on vital signs, it was found to reduce pain after cesarean section and it was not effective in reducing pain after cesarean section.

Although Reiki therapy has been proven to be effective in coping with many symptoms, studies on its effect on the level of fatigue and depression in the postpartum period are limited. It is predicted that Reiki will reduce the risk of depression by reducing the fatigue of women in the postpartum period and causing spiritual relaxation, due to its advantages such as not being an invasive procedure, ease of application and having no negative effects. For this reason, the research was conducted to evaluate the effect of Reiki therapy applied to women in the postpartum period on the risk of fatigue and postpartum depression.

ELIGIBILITY:
Inclusion Criteria:

* Participants were 18 years of age or older
* At least a primary school graduate
* Primiparous and multiparous, with a full-term (between 38-40 weeks) and healthy newborn
* Without any acute or chronic health problems, without communication problems that could answer the data collection tools used in the study
* Women who had not received body-mind therapy (yoga, reiki, meditation, etc.) in the last six months
* Women who agreed to participate to the research

Exclusion Criteria:

* Women who could not be contacted for the pre-test application on the 13th postpartum day
* Women who developed a health problem in themselves or/or their newborn
* Women who were diagnosed with a neuro-psychiatric disease
* Women who could not be reached by phone or SMS on the 13th and 14th postpartum days
* Women who wanted to leave the study voluntarily

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 85 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale for Fatigue (VAS-F) | two months
  Lee et al. (1990) and whose Turkish validity and reliability were determined by Yurtsever and Bedük (2003), the scale consists of 18 items. The scale is in the form of a 10 cm ruler with the most positive statements at one end and the most negative statements at the other end. The most positive expression of the fatigue sub-dimension is 0 and the most negative expression is 10. The most negative expression of the energy sub-dimension is 0 and the most positive expression is 10. The items of the fatigue sub-dimension are from the most positive to the most negative, and the items of the energy sub-dimension are from the most negative to the most positive. A high score of the fatigue sub-dimension and a low score of the energy sub-dimension indicate that the severity of fatigue is high. Evaluation of the scale is done by adding the total scores (0-180) obtained from the items. The scale does not have a cut-off point.
Edinburgh Postnatal Depression Scale (EPDS) | two months
  he scale prepared for screening purposes to determine the risk of depression in the postpartum period was developed by Cox et al. (1987), the scale is not intended to diagnose depression. EPDS consists of 10 items and is a 4-point Likert type. The answers to each question item are scored between 0-3 on a scale consisting of four options, the lowest score that can be obtained from the scale is 0 and the highest score is 30. In the evaluation, the 1st, 2nd, and 4th items are scored as 0, 1, 2, 3, and the 3rd, 5th, 6th, 7th, 8th, 9th, and 10th items are scored reversely as 3, 2, 1. is scored as 0. The total score of the scale is obtained by adding these item scores. The cut-off score of the scale is 12.5 and women whose total scale score is higher than the cut-off point are considered to be in the risk group. Turkish validity and reliability were determined by Aydin et al. (2004) Cronbach Alpha coefficient of the scale was found to be 0.76.

CONTACTS AND LOCATIONS:
Overall Officials: ILKNUR GOKSIN, PhD, Principal Investigator — Aksaray University
Locations (1):
- Aksaray University, Aksaray, Merkez, Turkey (Türkiye)